CLINICAL TRIAL: NCT03355274
Title: Application de l'oxymétrie Dynamique Pour le Diagnostic Des Syndromes de défilés Thoraco-brachiaux Systematic Transcutaneous Oxymetry Use in Thoracic Outlet Syndrom
Brief Title: Systematic Transcutaneous Oxymetry Use in Thoracic Outlet Syndrome
Acronym: STOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02554-49
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Transcutaneous Oximetry
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Blood Gas Monitoring, Transcutaneous

STUDY DESIGN:
Intervention Model Description: Patients with thoracic outlet syndrom (patients) Healthy asymptomatic patients (controls)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Patients suspected of thoracic outlet syndrome Transcutaneous oximetry during upper arm manoeuvers
  Interventions: Diagnostic Test: Transcutaneous Oximetry; Diagnostic Test: Photopletysmography; Other: Questionnaires of Quality of Life (QoL)
- controls (Sham Comparator): healthy asymptomatic subjects Transcutaneous oximetry during upper arm manoeuvers
  Interventions: Diagnostic Test: Transcutaneous Oximetry; Diagnostic Test: Photopletysmography; Other: Questionnaires of Quality of Life (QoL)

INTERVENTIONS:
Diagnostic Test: Transcutaneous Oximetry — The examination of transcutaneous Oximetry dynamic measurement with palmar face of both forearms during two consecutive maneuvers known as the "candlestick" (hands up).
Diagnostic Test: Photopletysmography — Maneuvers are repeted with the photoplestysmography sensors and in front of a Kinect camera.
Other: Questionnaires of Quality of Life (QoL) — Each subject complete 2 QoL questionnaires : Sf-12 (Short Form 12) and DASH (Disabilities of the Arm, Shoulder and Hand).

SUMMARY:
The measurement of the transcutaneous oxygen partial pressure (TCPO2) at exercise is, to our knowledge, the only method to estimate during the exercise the importance of ischemia segment of limb by segment of limb bilaterally and carry on. The diagnosis of thoracic outlet syndrome causing remains difficult and dependent operator in ultrasound because of the risk of false positive (loss of signal) or false negative (insufficient effort, inappropriate movement).

Our main hypothesis is the existence of significant measurable ischemia in the forearm by transcutaneous oximetry during the maneuvering of the "candlestick".

In the event of failure of this maneuver, the other maneuvers such as those of Wright, Roos, Tinel and Adson will be realized.

In this study we want to evaluate the possibility of using dynamic transcutaneous Oximetry as a tool for evaluating ischemia in case of suspicion of thoracic outlet syndrome causing.

DETAILED DESCRIPTION:
Patients referred for suspected thoracic outlet syndrome causing and healthy asymptomatic subjects will be included.

After signing the consent, the subject will have a clinical and paraclinical examination. Age, sex, height, weight, side of clinical symptomatology will be collected. Medical history current treatments will also be noted.

The examination of transcutaneous oximetry dynamic measurement with palmar face of both forearms during two consecutive maneuvers known as the "candlestick" (hands up). The most symptomatic arm value in patients and the dominant arm in the control group will be noted. In case of DROP between 0 and -25 mmHg, in addition to the maneuvering of the "candlestick", the other maneuvers such as those of Wright, Roos, Tinel and Adson will be realized.

The results of any additional examinations and / or pre- and post-operative consultations will be collected.

Subjects complete two Quality of Life questionnaires: the SF-12 (Short Form 12) and the DASH questionnaire (Disabilities of the Arm, Shoulder and Hand).

Added by an amendment : Photoplethysmography has already done its proofs to determine the thoracic outlet syndrome diagnotic. Combine with a camera Kinect, they should determine the angle of appearance of compression in the 3 dimensions of space.

ELIGIBILITY:
Inclusion Criteria:

* subjects referred for investigation of thoracic outlet syndrome causing
* Affiliation to the French National healthcare system
* French speaking patients
* Ability to stand still for half a minute

Exclusion Criteria:

* pregnancy
* inability to understand the study goal
* Patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Decrease from Rest of Oxygen Pressure (DROP) during manoeuvers in patients and controls. | inclusion
  Difference in DROP observed in the symptomatic arm of patients with suspected thoracic outlet syndrome compared to the dominant arm in controls

SECONDARY OUTCOMES:
Presence of stenosis or occlusion on angiography | 24 months
  The performance and cutoff of the DROP will be studied with the AUC (ROC curve) to predict a stenosis on angiography versus no stenosis in patients.
POsitive and negative DROP results | 24 months
  To determine the proportion of false positive and false negative results in controls using the cutoff determined in outcome 2
Angle of appearance of the compression observed on PPG | 24 months
  By combining the photopletysmography and a camera Kinect, it is possible to exactly determine the angle of appearance of the compression

CONTACTS AND LOCATIONS:
Overall Officials: Samir MD HENNI, PhD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France

REFERENCES:
- [Derived] Hersant J, Ramondou P, Guilleron C, Picquet J, Henni S, Abraham P. A pilot study of forearm microvascular impairment and pain while using a telephone. Microvasc Res. 2020 May;129:103963. doi: 10.1016/j.mvr.2019.103963. Epub 2019 Nov 29. PMID 31790665